CLINICAL TRIAL: NCT02691182
Title: Open-Label Extension Study to Evaluate the Long-Term Safety of Molindone Hydrochloride Extended-Release Tablets for the Treatment of Impulsive Aggression in Pediatric and Adolescent Subjects With Attention Deficit/Hyperactivity Disorder (ADHD) in Conjunction With Standard ADHD Treatment
Brief Title: Treatment of Impulsive Aggression in Subjects With ADHD in Conjunction With Standard ADHD Treatment (CHIME 4)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The program was shut down due to a lack of efficacy.
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810P304
Record Dates: First submitted 2016-02-02; First posted 2016-02-25 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (1):
- Open-label treatment with SPN-810 (Experimental): Subjects aged 6-17 years were treated with SPN-810 starting on day 1 with 18 mg/day. The clinician was able to adjust the dose of SPN-810 throughout the study based on subject's response and tolerability within the limits of 6 mg/day and 36 mg/day or, up to 54 mg/day for subjects with a body weight ≥ 30 kg.
  The subjects were given a choice of extending their participation in the study every 6-month period for up to 36 months
  Interventions: Drug: SPN-810

INTERVENTIONS:
Drug: SPN-810

SUMMARY:
Children between the ages of 6-12 years who are diagnosed with impulsive aggression comorbid with ADHD and have participated in the 810P301 or 810P302 study were invited to participate in this study. This was a Phase 3 open-label extension (OLE) study to collect long-term safety data on the use of SPN-810 in treating impulsive aggression in pediatric subjects with ADHD when taken in conjunction with standard ADHD treatment. After confirmation of eligibility, all subjects were treated with SPN-810. Subjects were given a choice to extend participation in this study every 6 months for up to 36 months.

DETAILED DESCRIPTION:
Study 810P304 is a multicenter, open-label, extension study aimed to assess safety of SPN-810 in the treatment of IA in patients aged 6-17 years with ADHD in conjunction with standard ADHD treatment.

The study has three phases: Optimization, Maintenance, and Taper. All subjects who complete the randomized, double-blind portion of study 810P301, 810P302, 810P503 or 810P204 will have the option to participate in the OLE study in which all subjects will receive active Study Medication (SM) treatment. Subjects who choose to participate in the OLE will receive blinded conversion medication kits at Visit 6 of the previous SPN-810 double-blind randomization study (810P301, 810P302) or at Visit 4 for subjects completing the 810P204 study. Subjects, who have completed the 810P503 study and, chose to participate in this study, will receive the blinded conversion card at Visit 7.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, who completed and converted from a satisfactory participation in the study 810P301, 810P302, 810P503 and 810P204 or discontinued early from the previous study during the maintenance phase and allowed to enroll only after consultation between the Investigator, the Medical Monitor and the Sponsor.
2. Medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs).
3. Existing diagnosis of ADHD, as described by DSM-5 and confirmed by the K-SADS PL 2013 from study 810P301 or 810P302 or by the MINI-KID from study 810P503 or 810P204.
4. Currently receiving monotherapy treatment with FDA-approved ADHD medication (stimulants and non-stimulants).
5. Weight of at least 20 kg.
6. Written Informed Consent obtained from the subject's parent or legally authorized representative (LAR), and written Informed Assent obtained from the subject if appropriate.

Exclusion Criteria:

1. Body Mass Index (BMI) in 99th percentile or above.
2. Clinically significant change in health status, safety concern or any other reason that, in the opinion of the Sponsor or the Investigator, would prevent the subject from participating in this study or successfully completing this study.
3. Pregnancy or refusal to practice contraception during the study (for female subjects of childbearing potential and sexually active males).
4. Current substance or alcohol use.
5. Suicidal thoughts or behaviors confirmed at Visit 7 for 810P301 or 810P302, Visit 8 for 810P503 or Visit 6 for 810P204 studies.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 491 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiera Ceresoli-Borroni, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (1):
- CNS Healthcare of Orlando, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- <18 mg SPN-810: Subjects treated with 6, 12 or 15 mg/day SPN-810.
- 18 mg to < 24 mg SPN-810: Subjects treated with 18 mg/day, or 21 mg/day SPN-810
- 24 mg to < 36 mg SPN-810: Subjects treated with 24, 27 or 30 mg/day SPN-810
- 36 mg to ≤54 mg SPN-810: Subjects treated with 36, 42, 45, 48 or 54 mg/day SPN-810
Period: Overall Study
Arm/Group | <18 mg SPN-810 | 18 mg to < 24 mg SPN-810 | 24 mg to < 36 mg SPN-810 | 36 mg to ≤54 mg SPN-810
Started (Number of subjects is based on the Safety Population, defined as all subjects who received at least 1 dose of study drug during the study.) | 38 | 159 | 131 | 163
Completed | 0 | 1 | 2 | 1
Not Completed | 38 | 158 | 129 | 162
Not completed — Withdrawal by Subject | 4 | 7 | 6 | 8
Not completed — Withdrawal by Parent/Guardian | 9 | 47 | 33 | 38
Not completed — Lost to Follow-up | 8 | 33 | 19 | 22
Not completed — Adverse Event | 3 | 10 | 10 | 11
Not completed — Physician Decision | 3 | 7 | 14 | 8
Not completed — Lack of Efficacy | 0 | 0 | 0 | 4
Not completed — Protocol Violation | 2 | 6 | 6 | 8
Not completed — Sponsor terminated study, SM non-compliance, Site closure, Subjects relocated or hospitalized. | 9 | 43 | 40 | 58
Not completed — Missing | 0 | 5 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Safety Population: Safety population is defined as all subjects who received at least 1 dose of study drug during the study.
Groups:
- <18 mg SPN-810: Subjects treated with 6,12 or 15 mg/day SPN-810
- 18 mg to <24 mg SPN-810: Subjects treated with 18 mg/day or 21 mg/day SPN-810
- 24 mg to <36 mg SPN-810: Subjects treated with 24, 27 or 30 mg/day SPN-810
- Total: Total of all reporting groups
Arm/Group | <18 mg SPN-810 | 18 mg to <24 mg SPN-810 | 24 mg to <36 mg SPN-810 | 36 mg to ≤54 mg SPN-810 | Total
Number analyzed (Participants) | 38 | 159 | 131 | 163 | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (1.78) | 9.3 (1.92) | 9.2 (1.91) | 9.9 (2.14) | 9.4 (2.02)
Age, Customized [Number; unit: participants]
  6-12 | 38 | 154 | 128 | 147 | 467
  12-17 | 0 | 5 | 3 | 16 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 34 | 29 | 32 | 104
  Male | 29 | 125 | 102 | 131 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 26 | 26 | 29 | 87
  Not Hispanic or Latino | 32 | 131 | 104 | 133 | 400
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 2 | 5
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 11 | 57 | 26 | 41 | 135
  White | 26 | 88 | 101 | 110 | 325
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 10 | 4 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Effect of SPN810 on Retrospective-Modified Overt Aggression Scale (R-MOAS) Total Score
Description: R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (VE, PH, PR, SE). For each open question in each area, the parent-rated the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: Verbal Incidents (VE)=1, Incidents Toward Other (PH) =4, Incidents Involving Property (PR)=2 and Incidents Directed Toward Self (SE)=3. Therefore, the sum of each area yields a maximum weighted score of 20 (VE), 120 (PH), 60 (PR), and 90 (SE). The total score is the sum of the four area scores or 0-290; the higher the score, the more severe the aggressive behavior is.
  The data represent the total score change from baseline at each visit for the duration of the study, a total of 60 months. The baseline score represents the total score at the last visit of each double-blind study.
Time Frame: 17-time points: Months 3 (V5), 6 (V6), 9 (V7), 12 (V8), 15 (V9), 18 (V10), 21 (V11), 24 (V12), 27 (V13), 30 (V14), 33 (V15), 36 (V16), 39 (V17), 42 (V18), 45 (V19), 48 (V20) and month 60 (Visit 24).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 18 mg to < 24 mg SPN-810: Subjects treated with 18 mg/day or 21 mg/day SPN-810
Arm/Group | <18 mg SPN-810 | 18 mg to < 24 mg SPN-810 | 24 mg to < 36 mg SPN-810 | 36 mg to ≤54 mg SPN-810
Number analyzed (Participants) | 38 | 159 | 131 | 163
score on a scale
  VE Score Month 3: number analyzed (Participants) | 26 | 123 | 114 | 138
  VE Score Month 3 | -7.1 (5.18) | -6.8 (5.57) | -5.5 (5.41) | -6.4 (5.84)
  PH Score Month 3: number analyzed (Participants) | 26 | 123 | 114 | 138
  PH Score Month 3 | -23.7 (17.41) | -18.5 (21.57) | -13.5 (17.28) | -16.9 (17.78)
  PR Score Month 3: number analyzed (Participants) | 26 | 123 | 114 | 138
  PR Score Month 3 | -16.1 (11.47) | -13.6 (13.48) | -9.9 (10.26) | -12.6 (11.90)
  SE Score Month 3: number analyzed (Participants) | 26 | 123 | 114 | 138
  SE Score Month 3 | -7.3 (10.15) | -6.3 (10.19) | -6.4 (9.42) | -5.3 (8.80)
  Total Score Month 3: number analyzed (Participants) | 26 | 123 | 114 | 138
  Total Score Month 3 | -54.1 (32.78) | -45.2 (40.50) | -35.2 (30.97) | -41.3 (34.02)
  VE Score Month 6: number analyzed (Participants) | 20 | 98 | 85 | 105
  VE Score Month 6 | -7.0 (4.62) | -5.4 (6.05) | -6.2 (4.93) | -5.9 (5.67)
  PH Score Month 6: number analyzed (Participants) | 20 | 98 | 85 | 105
  PH Score Month 6 | -23.6 (12.84) | -19.2 (24.44) | -16.1 (15.55) | -15.9 (17.62)
  PR Score Month 6: number analyzed (Participants) | 20 | 98 | 85 | 105
  PR Score Month 6 | -14.4 (10.54) | -12.5 (13.35) | -11.6 (11.27) | -11.8 (13.21)
  SE Score Month 6: number analyzed (Participants) | 20 | 98 | 85 | 105
  SE Score Month 6 | -7.2 (7.75) | -6.8 (10.29) | -7.5 (8.40) | -5.6 (8.78)
  Total Score Month 6: number analyzed (Participants) | 20 | 98 | 85 | 105
  Total Score Month 6 | -52.2 (26.54) | -44.0 (41.31) | -41.4 (28.50) | -39.2 (34.04)
  VE Score Month 9: number analyzed (Participants) | 19 | 74 | 68 | 85
  VE Score Month 9 | -6.4 (4.30) | -6.8 (5.03) | -6.5 (6.33) | -5.0 (5.97)
  PH Score Month 9: number analyzed (Participants) | 19 | 74 | 68 | 85
  PH Score Month 9 | -17.7 (15.79) | -22.6 (21.97) | -15.7 (16.05) | -13.7 (16.30)
  PR Score Month 9: number analyzed (Participants) | 19 | 74 | 68 | 85
  PR Score Month 9 | -13.9 (9.27) | -15.6 (11.85) | -11.7 (12.00) | -11.2 (12.98)
  SE Score Month 9: number analyzed (Participants) | 19 | 74 | 68 | 85
  SE Score Month 9 | -8.1 (8.72) | -7.1 (10.94) | -9.2 (8.92) | -6.6 (8.88)
  Total Score Month 9: number analyzed (Participants) | 19 | 74 | 68 | 85
  Total Score Month 9 | -46.1 (25.55) | -52.2 (39.56) | -43.2 (30.59) | -36.5 (33.44)
  VE Score Month 12: number analyzed (Participants) | 13 | 59 | 57 | 67
  VE Score Month 12 | -4.2 (5.57) | -6.6 (5.91) | -6.8 (4.81) | -5.9 (6.35)
  PH Score Month 12: number analyzed (Participants) | 13 | 59 | 57 | 67
  PH Score Month 12 | -11.1 (14.71) | -19.1 (19.43) | -18.2 (16.54) | -16.1 (18.18)
  PR Score Month 12: number analyzed (Participants) | 13 | 59 | 57 | 67
  PR Score Month 12 | -9.5 (12.63) | -14.4 (13.11) | -11.6 (10.50) | -11.8 (13.08)
  SE Score Month 12: number analyzed (Participants) | 13 | 59 | 57 | 67
  SE Score Month 12 | -2.8 (6.87) | -7.0 (11.80) | -8.5 (8.85) | -6.7 (8.40)
  Total Score Month 12: number analyzed (Participants) | 13 | 59 | 57 | 67
  Total Score Month 12 | -27.6 (28.46) | -47.0 (40.33) | -45.2 (28.69) | -40.4 (34.34)
  VE Score Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  VE Score Month 15 | -5.5 (3.87) | -7.2 (6.26) | -7.2 (4.91) | -6.2 (6.05)
  PH Score Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  PH Score Month 15 | -14.4 (15.11) | -20.7 (19.65) | -17.3 (14.86) | -16.5 (18.43)
  PR Score Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  PR Score Month 15 | -13.4 (10.59) | -16.5 (12.78) | -13.2 (11.45) | -13.5 (12.34)
  SE Score Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  SE Score Month 15 | -4.5 (5.87) | -6.3 (12.96) | -9.9 (8.84) | -6.7 (8.15)
  Total Score Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  Total Score Month 15 | -37.8 (26.08) | -50.7 (43.31) | -47.6 (26.68) | -42.9 (33.47)
  VE Score Month 18: number analyzed (Participants) | 8 | 39 | 37 | 42
  VE Score Month 18 | -5.8 (7.03) | -6.7 (6.49) | -7.0 (4.77) | -6.9 (5.79)
  PH Score Month 18: number analyzed (Participants) | 8 | 39 | 37 | 42
  PH Score Month 18 | -15.5 (15.03) | -24.0 (20.50) | -16.9 (15.12) | -19.9 (19.78)
  PR Score Month 18: number analyzed (Participants) | 8 | 39 | 37 | 42
  PR Score Month 18 | -17.3 (10.36) | -17.5 (13.01) | -13.9 (10.45) | -15.0 (10.45)
  SE Score Month 18: number analyzed (Participants) | 8 | 39 | 37 | 42
  SE Score Month 18 | -1.5 (4.24) | -7.8 (12.94) | -9.8 (8.74) | -6.1 (9.38)
  Total Score Month 18: number analyzed (Participants) | 8 | 39 | 37 | 42
  Total Score Month 18 | -40.0 (30.85) | -56.0 (42.08) | -47.6 (25.64) | -47.8 (36.62)
  VE Score Month 21: number analyzed (Participants) | 6 | 33 | 29 | 36
  VE Score Month 21 | -7.0 (4.69) | -6.9 (6.84) | -7.9 (5.71) | -6.7 (5.66)
  PH Score Month 21: number analyzed (Participants) | 6 | 33 | 29 | 36
  PH Score Month 21 | -20.0 (8.00) | -22.7 (21.11) | -18.3 (14.44) | -19.9 (18.08)
  PR Score Month 21: number analyzed (Participants) | 6 | 33 | 29 | 36
  PR Score Month 21 | -11.7 (10.84) | -18.7 (13.19) | -15.2 (11.67) | -13.4 (12.71)
  SE Score Month 21: number analyzed (Participants) | 6 | 33 | 29 | 36
  SE Score Month 21 | -2.5 (3.99) | -10.0 (13.05) | -9.9 (9.95) | -7.2 (8.03)
  Total Score Month 21: number analyzed (Participants) | 6 | 33 | 29 | 36
  Total Score Month 21 | -41.2 (12.80) | -58.3 (45.11) | -51.4 (27.49) | -47.1 (34.49)
  VE Score Month 24: number analyzed (Participants) | 6 | 31 | 22 | 33
  VE Score Month 24 | -6.0 (5.66) | -7.5 (5.18) | -8.3 (5.50) | -5.5 (5.55)
  PH Score Month 24: number analyzed (Participants) | 6 | 31 | 22 | 33
  PH Score Month 24 | -16.7 (13.25) | -24.3 (19.04) | -19.6 (15.95) | -17.7 (18.19)
  PR Score Month 24: number analyzed (Participants) | 6 | 31 | 22 | 33
  PR Score Month 24 | -13.3 (10.25) | -19.2 (9.87) | -14.2 (11.82) | -13.3 (9.24)
  SE Score Month 24: number analyzed (Participants) | 6 | 31 | 22 | 33
  SE Score Month 24 | 1.5 (6.50) | -8.9 (12.01) | -8.9 (8.10) | -6.0 (8.68)
  Total Score Month 24: number analyzed (Participants) | 6 | 31 | 22 | 33
  Total Score Month 24 | -34.5 (27.24) | -59.9 (34.30) | -51.0 (27.96) | -42.6 (33.62)
  VE Score Month 27: number analyzed (Participants) | 5 | 25 | 17 | 23
  VE Score Month 27 | -6.4 (6.80) | -7.6 (5.69) | -8.8 (5.51) | -6.7 (3.79)
  PH Score Month 27: number analyzed (Participants) | 5 | 25 | 17 | 23
  PH Score Month 27 | -19.2 (15.07) | -23.5 (19.26) | -17.4 (18.65) | -24.7 (19.17)
  PR Score Month 27: number analyzed (Participants) | 5 | 25 | 17 | 23
  PR Score Month 27 | -11.6 (7.92) | -18.2 (10.48) | -16.5 (11.91) | -14.5 (11.25)
  SE Score Month 27: number analyzed (Participants) | 5 | 25 | 17 | 23
  SE Score Month 27 | 1.8 (5.85) | -10.3 (13.75) | -9.0 (7.65) | -5.9 (7.86)
  Total Score Month 27: number analyzed (Participants) | 5 | 25 | 17 | 23
  Total Score Month 27 | -35.4 (28.79) | -59.6 (37.18) | -51.6 (32.26) | -51.8 (29.04)
  VE Score Month 30: number analyzed (Participants) | 4 | 21 | 12 | 20
  VE Score Month 30 | -10.0 (4.24) | -8.3 (5.79) | -8.8 (5.34) | -6.8 (4.97)
  PH Score Month 30: number analyzed (Participants) | 4 | 21 | 12 | 20
  PH Score Month 30 | -17.0 (17.70) | -19.6 (20.55) | -23.0 (16.81) | -22.2 (16.34)
  PR Score Month 30: number analyzed (Participants) | 4 | 21 | 12 | 20
  PR Score Month 30 | -14.5 (9.85) | -17.7 (10.32) | -16.7 (14.51) | -13.5 (13.45)
  SE Score Month 30: number analyzed (Participants) | 4 | 21 | 12 | 20
  SE Score Month 30 | -2.3 (2.87) | -8.9 (13.70) | -6.8 (9.15) | -4.9 (9.60)
  Total Score Month 30: number analyzed (Participants) | 4 | 21 | 12 | 20
  Total Score Month 30 | -43.8 (30.91) | -54.5 (39.26) | -55.3 (29.39) | -47.7 (31.41)
  VE Score Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  VE Score Month 33 | -8.5 (4.95) | -6.8 (3.12) | -11.0 (4.32) | -5.7 (5.99)
  PH Score Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  PH Score Month 33 | -24.0 (16.97) | -11.5 (23.07) | -42.0 (13.66) | -15.7 (14.33)
  PR Score Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  PR Score Month 33 | -14.0 (11.31) | -15.7 (12.46) | -18.0 (17.05) | -12.0 (8.41)
  SE Score Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  SE Score Month 33 | 0.0 (0.00) | -5.4 (8.58) | -8.3 (7.50) | -3.0 (11.16)
  Total Score Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  Total Score Month 33 | -46.5 (33.23) | -39.4 (34.32) | -79.3 (37.29) | -36.4 (33.14)
  VE Score Month 36: number analyzed (Participants) | 1 | 12 | 3 | 13
  VE Score Month 36 | -6.0 | -7.3 (3.65) | -7.7 (5.03) | -7.9 (7.06)
  PH Score Month 36: number analyzed (Participants) | 1 | 12 | 3 | 13
  PH Score Month 36 | -4.0 | -14.3 (9.26) | -30.7 (6.11) | -26.5 (16.13)
  PR Score Month 36: number analyzed (Participants) | 1 | 12 | 3 | 13
  PR Score Month 36 | -8.0 | -17.2 (6.41) | -12.0 (6.00) | -17.1 (9.30)
  SE Score Month 36: number analyzed (Participants) | 1 | 12 | 3 | 13
  SE Score Month 36 | 0.0 | -8.8 (9.78) | -4.0 (6.24) | -5.5 (6.91)
  Total Score Month 36: number analyzed (Participants) | 1 | 12 | 3 | 13
  Total Score Month 36 | -18.0 | -47.5 (12.53) | -54.3 (15.04) | -57.0 (29.94)
  VE Score Month 39: number analyzed (Participants) | 1 | 7 | 2 | 11
  VE Score Month 39 | 4.0 | -5.3 (4.39) | -0.5 (10.61) | -7.5 (3.50)
  PH Score Month 39: number analyzed (Participants) | 1 | 7 | 2 | 11
  PH Score Month 39 | -12.0 | -13.1 (7.90) | -6.0 (42.43) | -22.5 (14.78)
  PR Score Month 39: number analyzed (Participants) | 1 | 7 | 2 | 10
  PR Score Month 39 | -4.0 | -15.4 (5.97) | -7.0 (15.56) | -16.6 (10.02)
  SE Score Month 39: number analyzed (Participants) | 1 | 7 | 2 | 10
  SE Score Month 39 | 0.0 | -7.7 (5.71) | 4.5 (6.36) | -3.9 (9.06)
  Total Score Month 39: number analyzed (Participants) | 1 | 7 | 2 | 11
  Total Score Month 39 | -12.0 | -41.6 (13.18) | -9.0 (31.11) | -51.6 (27.62)
  VE Score Month 42: number analyzed (Participants) | 0 | 1 | 2 | 7
  VE Score Month 42 |  | -7.0 | -9.0 (7.07) | -8.9 (5.37)
  PH Score Month 42: number analyzed (Participants) | 0 | 1 | 2 | 7
  PH Score Month 42 |  | -12.0 | -14.0 (19.80) | -27.4 (13.55)
  PR Score Month 42: number analyzed (Participants) | 0 | 1 | 2 | 7
  PR Score Month 42 |  | -18.0 | -7.0 (7.07) | -15.1 (13.85)
  SE Score Month 42: number analyzed (Participants) | 0 | 1 | 2 | 7
  SE Score Month 42 |  | -3.0 | -3.0 (4.24) | -5.6 (8.20)
  Total Score Month 42: number analyzed (Participants) | 0 | 1 | 2 | 7
  Total Score Month 42 |  | -40.0 | -33.0 (15.56) | -57.0 (32.17)
  VE Score Month 45: number analyzed (Participants) | 0 | 1 | 0 | 3
  VE Score Month 45 |  | -7.0 |  | -8.3 (2.08)
  PH Score Month 45: number analyzed (Participants) | 0 | 1 | 0 | 3
  PH Score Month 45 |  | -8.0 |  | -24.0 (16.00)
  PR Score Month 45: number analyzed (Participants) | 0 | 1 | 0 | 3
  PR Score Month 45 |  | -14.0 |  | -14.7 (7.57)
  SE Score Month 45: number analyzed (Participants) | 0 | 1 | 0 | 3
  SE Score Month 45 |  | -18.0 |  | -2.0 (9.17)
  Total Score Month 45: number analyzed (Participants) | 0 | 1 | 0 | 3
  Total Score Month 45 |  | -47.0 |  | -49.0 (22.07)
  VE Score Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  VE Score Month 48 |  |  |  | -9.0
  PH Score Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  PH Score Month 48 |  |  |  | -28.0
  PR Score Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  PR Score Month 48 |  |  |  | -6.0
  SE Score Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  SE Score Month 48 |  |  |  | -12.0
  Total Score Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  Total Score Month 48 |  |  |  | -55.0
  VE Score Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  VE Score Month 60 |  |  | -10.0 | -12.0
  PH Score Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  PH Score Month 60 |  |  | 12.0 | -12.0
  PR Score Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  PR Score Month 60 |  |  | -12.0 | -12.0
  SE Score Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  SE Score Month 60 |  |  | 3.0 | -6.0
  Total Score Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  Total Score Month 60 |  |  | -7.0 | -42.0

2. Primary Outcome: Effect of SPN810 on Impulsive Aggression (IA) Measured by Clinical Global Impression - Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of the severity of IA behaviors. CGI-S was evaluated by the Investigator at each visit on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill.
  Data represent the change from baseline to each visit during the study. The baseline score represents the total score at the last visit of each double-blind study.
Time Frame: 20-time points: Week 2 (V2), Week 4 (V3), Week 8 (V4), Months 3 (V5), 6 (V6), 9 (V7), 12 (V8), 15 (V9),18 (V10), 21 (V11), 24 (V12), 27 (V13), 30 (V14), 33 (V15), 36 (V16), 39 (V17), 42 (V18), 45 (V19), 48 (V20) and month 60 (Visit 24).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- <18 mg SPN-810: Subjects treated 6, 12 or 15 mg/day SPN-810
- 24 to < 36 mg SPN-810: Subjects treated with 24, 27 or 30 mg/day SPN-810
Arm/Group | <18 mg SPN-810 | 18 mg to < 24 mg SPN-810 | 24 to < 36 mg SPN-810 | 36 mg to ≤54 mg SPN-810
Number analyzed (Participants) | 38 | 159 | 131 | 163
score on a scale
  Week 2: number analyzed (Participants) | 38 | 147 | 131 | 162
  Week 2 | -1.2 (1.33) | -1.8 (1.13) | -1.0 (0.94) | -1.0 (0.95)
  Week 4: number analyzed (Participants) | 35 | 141 | 128 | 162
  Week 4 | -1.6 (1.26) | -2.1 (1.10) | -1.2 (1.12) | -1.3 (1.06)
  Week 8: number analyzed (Participants) | 29 | 135 | 120 | 150
  Week 8 | -2.0 (1.20) | -2.1 (1.18) | -1.4 (1.13) | -1.5 (1.02)
  Month 3: number analyzed (Participants) | 26 | 122 | 114 | 138
  Month 3 | -1.9 (1.37) | -2.2 (1.08) | -1.5 (1.15) | -1.6 (0.98)
  Month 6: number analyzed (Participants) | 21 | 97 | 84 | 104
  Month 6 | -2.0 (0.95) | -2.2 (1.07) | -1.5 (0.95) | -1.8 (0.95)
  Month 9: number analyzed (Participants) | 18 | 72 | 68 | 84
  Month 9 | -1.9 (0.90) | -2.2 (1.02) | -1.8 (0.92) | -1.8 (0.97)
  Month 12: number analyzed (Participants) | 13 | 59 | 57 | 68
  Month 12 | -1.5 (1.13) | -2.3 (0.96) | -2.0 (1.01) | -1.8 (1.03)
  Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  Month 15 | -1.7 (1.25) | -2.3 (0.93) | -1.9 (0.90) | -1.8 (0.97)
  Month 18: number analyzed (Participants) | 8 | 39 | 38 | 42
  Month 18 | -1.5 (1.51) | -2.1 (1.03) | -2.0 (1.08) | -2.0 (0.90)
  Month 21: number analyzed (Participants) | 6 | 33 | 28 | 37
  Month 21 | -2.3 (1.03) | -2.2 (1.01) | -1.9 (1.03) | -1.9 (0.92)
  Month 24: number analyzed (Participants) | 6 | 32 | 22 | 32
  Month 24 | -2.5 (1.05) | -2.3 (0.89) | -2.1 (1.13) | -1.9 (0.98)
  Month 27: number analyzed (Participants) | 5 | 25 | 17 | 21
  Month 27 | -1.8 (1.48) | -2.2 (0.87) | -1.9 (1.03) | -2.0 (0.95)
  Month 30: number analyzed (Participants) | 4 | 20 | 12 | 20
  Month 30 | -2.0 (1.83) | -2.4 (0.88) | -2.0 (1.13) | -2.2 (0.99)
  Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  Month 33 | -3.5 (0.71) | -2.3 (1.03) | -2.8 (1.71) | -1.8 (0.89)
  Month 36: number analyzed (Participants) | 1 | 12 | 3 | 14
  Month 36 | -4.0 | -2.6 (0.79) | -1.7 (0.58) | -1.9 (0.73)
  Month 39: number analyzed (Participants) | 1 | 7 | 2 | 11
  Month 39 | -4.0 | -2.7 (0.95) | -1.5 (0.71) | -2.1 (0.70)
  Month 42: number analyzed (Participants) | 0 | 2 | 2 | 7
  Month 42 |  | -3.0 (0.00) | -2.0 (0.00) | -2.0 (1.15)
  Month 45: number analyzed (Participants) | 0 | 1 | 0 | 2
  Month 45 |  | -4.0 |  | -2.0 (0.00)
  Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  Month 48 |  |  |  | -3.0
  Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  Month 60 |  |  | -1.0 | -3.0

3. Primary Outcome: Effect of SPN810 on Impulsive Aggression (IA) Measured by Clinical Global Impression - Improvement Scale (CGI-I)
Description: The Clinical Global Impression - Improvement Scale (CGI-I) is a clinician's assessment of how much the IA behaviors have improved or worsened relative to a baseline state at the beginning of treatment. CGI-I was evaluated by the Investigator at each visit on a 7-point scale with 1=Very much improved, 2= Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse.
  Data represent the score at each visit during the study.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 18 mg to < 24mg SPN-810: Subjects treated with 18 mg/day or 21 mg/day SPN-810
- 24 to <36 mg SPN-810: Subjects treated with 24, 27 or 30 mg/day SPN-810
- 36 to ≤54 mg SPN-810: Subjects treated with 36, 42, 45, 48 or 54 mg/day SPN-810
Arm/Group | <18 mg SPN-810 | 18 mg to < 24mg SPN-810 | 24 to <36 mg SPN-810 | 36 to ≤54 mg SPN-810
Number analyzed (Participants) | 38 | 159 | 131 | 163
score on a scale
  Week 2: number analyzed (Participants) | 38 | 147 | 131 | 163
  Week 2 | 2.7 (1.25) | 2.1 (0.96) | 2.9 (1.19) | 2.9 (0.98)
  Week 4: number analyzed (Participants) | 35 | 141 | 128 | 163
  Week 4 | 2.1 (1.00) | 1.9 (0.94) | 2.6 (1.18) | 2.7 (1.02)
  Week 8: number analyzed (Participants) | 29 | 135 | 120 | 151
  Week 8 | 1.9 (0.80) | 1.9 (1.05) | 2.4 (0.97) | 2.5 (1.05)
  Month 3: number analyzed (Participants) | 26 | 122 | 114 | 139
  Month 3 | 1.9 (0.98) | 1.8 (0.84) | 2.4 (1.11) | 2.3 (1.06)
  Month 6: number analyzed (Participants) | 21 | 97 | 85 | 105
  Month 6 | 1.7 (0.66) | 1.7 (0.78) | 2.2 (1.13) | 2.2 (1.02)
  Month 9: number analyzed (Participants) | 18 | 73 | 68 | 85
  Month 9 | 1.8 (0.65) | 1.7 (0.69) | 2.0 (0.80) | 2.1 (0.91)
  Month 12: number analyzed (Participants) | 13 | 59 | 57 | 68
  Month 12 | 2.5 (1.33) | 1.8 (1.10) | 1.9 (0.80) | 2.1 (0.92)
  Month 15: number analyzed (Participants) | 10 | 47 | 48 | 56
  Month 15 | 2.3 (1.77) | 1.8 (1.11) | 2.0 (0.76) | 2.1 (0.80)
  Month 18: number analyzed (Participants) | 7 | 39 | 38 | 42
  Month 18 | 2.6 (2.07) | 1.9 (1.11) | 1.9 (0.71) | 1.9 (0.64)
  Month 21: number analyzed (Participants) | 6 | 33 | 28 | 37
  Month 21 | 1.5 (0.55) | 1.7 (0.67) | 2.0 (0.77) | 1.9 (0.76)
  Month 24: number analyzed (Participants) | 6 | 32 | 22 | 32
  Month 24 | 1.2 (0.41) | 1.7 (0.60) | 2.0 (0.72) | 1.8 (0.98)
  Month 27: number analyzed (Participants) | 5 | 25 | 17 | 21
  Month 27 | 2.4 (1.52) | 1.6 (0.49) | 1.7 (0.69) | 1.9 (1.00)
  Month 30: number analyzed (Participants) | 4 | 20 | 12 | 20
  Month 30 | 2.3 (1.89) | 1.5 (0.51) | 1.8 (0.75) | 1.9 (1.21)
  Month 33: number analyzed (Participants) | 2 | 15 | 4 | 14
  Month 33 | 1.0 (0.00) | 1.5 (0.64) | 1.8 (0.96) | 1.9 (0.66)
  Month 36: number analyzed (Participants) | 1 | 12 | 3 | 14
  Month 36 | 1.0 | 1.5 (0.52) | 2.3 (0.58) | 1.9 (0.73)
  Month 39: number analyzed (Participants) | 1 | 7 | 2 | 11
  Month 39 | 1.0 | 1.3 (0.49) | 2.5 (0.71) | 1.5 (0.52)
  Month 42: number analyzed (Participants) | 0 | 2 | 2 | 7
  Month 42 |  | 1.5 (0.71) | 2.0 (0.00) | 1.7 (1.11)
  Month 45: number analyzed (Participants) | 0 | 1 | 0 | 2
  Month 45 |  | 1.0 |  | 1.5 (0.71)
  Month 48: number analyzed (Participants) | 0 | 0 | 0 | 1
  Month 48 |  |  |  | 1.0
  Month 60: number analyzed (Participants) | 0 | 0 | 1 | 1
  Month 60 |  |  | 3.0 | 1.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each study visit: Visit 1 (last visit in the double-blind study), weeks 2,4 and 8, and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48 and 60 (months).
Description: Adverse events reporting pertains to the Safety Population, defined as all subjects who received at least 1 dose of study drug during the study.
Arm/Group | <18 mg SPN-810 | 18 mg to < 24 mg SPN-810 | 24 mg to < 36 mg SPN-810 | 36 mg to ≤54 mg SPN-810
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/159 | 0/131 | 0/163
Serious Adverse Events (participants affected / at risk) | 3/38 | 5/159 | 5/131 | 9/163
Other Adverse Events (participants affected / at risk) | 18/38 | 56/159 | 56/131 | 66/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | <18 mg SPN-810 (N=38) | 18 mg to < 24 mg SPN-810 (N=159) | 24 mg to < 36 mg SPN-810 (N=131) | 36 mg to ≤54 mg SPN-810 (N=163)
Suicidal Ideation (Psychiatric disorders) | 0 | 2 (2) | 3 (3) | 2 (2)
Aggression (Psychiatric disorders) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Oppositional Defiant Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious Mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain Mass (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | <18 mg SPN-810 (N=38) | 18 mg to < 24 mg SPN-810 (N=159) | 24 mg to < 36 mg SPN-810 (N=131) | 36 mg to ≤54 mg SPN-810 (N=163)
Nasopharyngitis (Infections and infestations) | 1 (1) | 10 (10) | 11 (13) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 14 (17) | 7 (13) | 12 (15)
Influenza (Infections and infestations) | 2 (3) | 5 (5) | 5 (5) | 7 (7)
Gastroenteritis (Infections and infestations) | 2 (2) | 6 (6) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 5 (5) | 13 (13) | 20 (21)
Blood prolactin increased (Investigations) | 1 (1) | 9 (11) | 10 (13) | 8 (8)
Tic (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 9 (12) | 11 (14) | 12 (20)
Somnolence (Nervous system disorders) | 3 (3) | 3 (4) | 6 (7) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (9) | 11 (13) | 9 (11)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 6 (6) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 7 (8) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02691182/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT02691182/SAP_001.pdf